CLINICAL TRIAL: NCT04703335
Title: Pilot Clinical Trial - Comparative Study of Two Material Concentration of OD-141309 With Controls When Used as a Preoperative Skin Disinfection Preparation.
Brief Title: Pilot Clinical Trial - Comparative Study of Two Material Concentration of OD-141309
Acronym: Odysseus-01
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zaycor Healthcare Corp (Industry)
Collaborators: BioScience Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OD-01-SSI-141309
Record Dates: First submitted 2021-01-05; First posted 2021-01-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Non-inferiority and Persistence (Experimental): Evaluate the antimicrobial efficacy of two concentrations of one patient preoperative skin preparation product compared to a positive control (2.0% chlorhexidine gluconate) and negative control (physiological saline 0.9% solution).
  Interventions: Drug: Antimicrobial efficacy of gel ZHCK4 as a patient preoperative skin preparation

INTERVENTIONS:
Drug: Antimicrobial efficacy of gel ZHCK4 as a patient preoperative skin preparation — Evaluate the antimicrobial efficacy of two concentrations of one patient preoperative skin preparation product compared to a positive control (2.0% chlorhexidine gluconate) and negative control (physiological saline 0.9% solution). Following a 14-day restriction period, subjects will be sampled for baseline, 10-minutes, 6-hours, and 24-hours microbial reduction evaluations post-product application. Subjects will not be sequestered for the 6-hour or 24-hour evaluations. Test day baseline criteria will be set at: abdomen: ≥ 3.0 log10 CFU/cm2, and inguen: ≥ 5.0 log10 CFU/cm2.

SUMMARY:
A sufficient number of subjects will be entered into testing to complete 42 subjects per each of the 2 test and 2 control configurations. A total of 84 subjects, testing bi-laterally (168 abdomen and groin sites in total completed, 42 abdomen and groin sites per each test and control material) will be evaluated using the standardized ASTM E1173 test method. Following a 14-day restriction period, subjects will be sampled for baseline, 10 minutes, 6 hours, and 24 hours post application (subjects will not be sequestered) for microbial reduction evaluations. Test day baseline criteria will be set at: abdomen: ≥ 3.0 log10 CFU/cm2, and groin: ≥ 5.0 log10 CFU/cm2.

DETAILED DESCRIPTION:
At least 84 subjects will be treated bilaterally with two of the four test materials (Test Product #1, Test Product #2, Positive Control, and Negative Control), one per each side of the abdomen and inguinal test sites. Subjects will be required to complete a 14-day pretest conditioning period. Subjects will complete a 2-day test period, during which time subjects' sites will be treated with the test materials and samples taken following treatment. The Cylinder Sampling Technique will be performed for baseline and for sampling 10-minutes, 6-hours, and 24-hours post-test material-application on Test Days.

The effectiveness criteria are that the log10 recoveries of the two test products (1% and 1.5%) are non-inferior to the Positive Control (2.0% chlorhexidine gluconate) with a 0.5 margin (log10 scale) per square centimeter on the abdominal and inguinal sites within 10 minutes after drying. The determination of non-inferiority will be based on the upper bounds of the 95% confidence interval being equal to or less than 0.5. Superiority will not be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be of either sex, at least 18 years of age and no more than 65 years of age, and of any race.
* Subjects must be able to read and understand English.
* Subjects must read and sign an Informed Consent Form, List of Restricted Products Form, and Allowed and Restricted Products for Hand Cleaning During Coronavirus Disease 2019 (COVID-19) Pandemic Form prior to participating in the study, as well as have an Authorization to Use and Disclose Protected Health Information Form on file at the testing facility.
* Subjects must be in good general health and have no medical diagnosis of a physical condition, such as a current or recent severe illness, medicated or uncontrolled diabetes, hepatitis B, hepatitis C, an organ transplant, mitral valve prolapse with heart murmur, fibromyalgia, ulcerative colitis, Crohn's disease, asthma, lung disease, liver disease, kidney disease, heart disease, hypertension, an immunocompromised condition such as AIDS (or HIV positive), lupus, medicated multiple sclerosis and must not have a history of smoking or vaping in the past 2 years.
* Subjects will have test sites on the skin of the abdomen and/or inguinal free of injury and in good condition (no active skin rashes, excessive freckling, moles, scratches, breaks in the skin, etc.) and have no currently active skin diseases or skin conditions (for example, contact dermatitis, psoriasis or eczema) that may compromise subject safety or study integrity.
* Subjects must have skin within 6 inches of the test sites that is free of tattoos, dermatoses, abrasions, cuts, lesions or other skin disorders. Subjects with tattoos, scars, active skin rashes, or breaks in the skin of test sites, skin blemishes, such as dry scabs or warts, may be admitted at the discretion of the Principal Investigator, Subinvestigators, or Consulting Physicians.
* Subjects must be able to lay on their backs with one leg bent to expose inguinal test site for approximately 20 minutes

Exclusion Criteria:

* Known allergies to vinyl, latex (rubber), alcohols, metals, tapes or adhesives, inks, sunscreens, deodorants, laundry detergents, topically applied fragrances, cleansers, or to common antibacterial agents found in soaps or lotions, particularly chlorhexidine gluconate, perillyl alcohol or isopropanol.
* Have experienced hives (raised welts) as a reaction to anything that contacted the skin with the exception of items that cause hives as a reaction to the general population (e.g. poison oak and poison ivy).
* Use of systemic or topical antibiotic medications.
* Use of systemic or topical steroids, other than for contraception, hormone therapy, post-menopausal indications. This includes steroid medications used to treat asthma. Note: topically applied hormonal steroids used for post-menopausal reasons must not get on the test sites.
* Any type of port (or portacath) or Peripherally Inserted Central Catheter (PICC).
* Pregnancy, plans to become pregnant or impregnate a sexual partner within the pre-test and test period of the study, or nursing a child. Female subjects must have a negative urine pregnancy test documented before treatment with test materials.
* Current participation or participation in a clinical study in the 14 days prior to the first lab visit.
* Any medical condition or use of any medications that, in the opinion of the Principal Investigator or Consulting Physicians, would preclude participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Antimicrobial efficacy | 10-minutes
  A primary efficacy variable for this study is the immediate antimicrobial effect at 10-minutes post-application of the change on measurement of two-test products against a positive control on the skin flora. The effectiveness criteria are that the log10 recoveries of the two test products (1% and 1.5%) are non-inferior to the Positive Control (2.0% chlorhexidine gluconate) with a 0.5 margin (log10 scale) per square centimeter on the abdominal and inguinal sites within 10 minutes after drying. The determination of non-inferiority will be based on a log10 multiple linear regression model. The Average Treatment Effect (ATE) is the mean difference of the test and the positive control products used in performing a non-inferiority statistic.

SECONDARY OUTCOMES:
Persistence of Antimicrobial Effect | 6-hours
  The log10 recoveries of the change in baseline measurements on skin flora by two test products (1% and 1.5%) must show to be superior to the Negative Control with a 1.2 margin (log10 scale) per square centimeter on the abdominal and inguinal sites within 10 minutes after drying. The determination of superiority will be based on a log10 multiple linear regression model. The Average Treatment Effect (ATE) is the mean difference of the test and the negative control products used in performing a superiority statistic.
  To demonstrate persistence for the test materials, the 6-hour post-treatment measurement should be lower than or equal to the baseline measurement for 100 percent of the subjects on the abdominal and inguinal sites.